CLINICAL TRIAL: NCT04893746
Title: Lactobacillus Plantarum TWK10 Improves Muscle Mass and Functional Performance in Frail Older Adults: A Randomized, Double-Blind Clinical Trial
Brief Title: TWK10 Improves Muscle Mass and Functional Performance in Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Synbio Tech Inc. (Industry)
Responsible Party: Principal Investigator, Chi-Chang Huang, PI, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00003
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Frail Elderly Syndrome; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin
- TWK10-L (Experimental): Low dose
  Interventions: Dietary Supplement: Lactobacillus plantarum TWK10-L
- TWK10-H (Experimental): High dose
  Interventions: Dietary Supplement: Lactobacillus plantarum TWK10-H

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum TWK10-L — Low dose: 2x1010 CFU/day
  Arms: TWK10-L
Dietary Supplement: Maltodextrin — 0x1010 CFU/day
  Arms: Placebo
Dietary Supplement: Lactobacillus plantarum TWK10-H — High dose: 6x1010 CFU/day
  Arms: TWK10-H

SUMMARY:
To explore the effect of "Lactobacillus plantarum TWK10 (hereinafter referred to as TWK10)" produced by synbiotech Biotechnology Co., Ltd. on alleviating and improving the aging and debilitating diseases of the elderly. Methods: It is expected to recruit 55-85-year-old senior citizens, who are assessed by the Clinical Frailty Scale (CFS) as debilitating disease grades 1 to 4 as the experimental subjects of this study. All subjects were divided into three groups according to the principle of balance order of frailty grades, namely (1) placebo group (Placebo group, average 77.4 years old), (2) supplement TWK10 probiotic 2x1010 CFU/day dose group (TWK10-L) Group, average 77.1 years old), (3) supplemented with TWK10 probiotic 6x1010 CFU/day dose group (TWK10-H group, average 79.0 years old). The experiment was supplemented for 24 consecutive weeks, and before supplementation, 6 weeks, 12 weeks, 18 weeks, the whole body composition and bone density test, as well as the functional fitness test were carried out in sequence. The items include: 3 meters walking ( Balance and gait assessment), 10-meter walking, 30-second sit-ups, and changes in the maximum grip strength of the left and right hands. Results: The experimental data showed that in the functional test, supplementing the TWK10-H group significantly improved the 3m gait balance, 10m walking, and lower limb muscle strength (30-second sit-ups) in the functional test. In terms of body composition and bone density, TWK10-H can significantly increase relative muscle mass after 18 weeks of supplementation. Conclusion: This study confirmed that supplementation of Lactobacillus plantarum TWK10 for 18 consecutive weeks can significantly promote the improvement of functional tests for the elderly, such as: 3m gait balance, 10m walking, lower limb muscle strength and grip strength, and can maintain and improve muscle mass. It has the effect of improving the frailty and muscle loss of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* The clinical frailty scale (Clinical Frailty Scale, CFS) assessed as frailty grade 1~4.

Exclusion Criteria:

* Diagnosed by the attending physician and confirmed that there is no stroke, hypertension patients and no exercise contraindications
* Can't sit to stand independently
* long-term antibiotics.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Grip strength | every 6 weeks
  Use the armed grip machine (T.K.K.5401, Takei Scientific Instruments Co.,Ltd, Niigata, Japan) to measure, hold each of the left and right hands three times until they are weak, and record the maximum value
3 meter walk | every 6 weeks
  Use a pyramid, a chair, and a measuring tape to measure a distance of three meters, and ask the subject to stand up from the chair, go around the pyramid and sit down, and record the time
30 second up to sit | every 6 weeks
  Use a stopwatch to record the number of times get up from the chair in 30 seconds
10 meter walk | every 6 weeks
  Use a pyramid and a measuring tape to measure a distance of ten meters, and ask the subject to stand up from the chair, go around the pyramid and sit down, and record the time
muscle mass | every 6 weeks
  Use dual-energy X-ray absorptiometry, DXA (Lunar iDXA, GE Healthcare, IL, USA) for no-entry measurement to determine muscle mass
fat percentage | every 6 weeks
  Use dual-energy X-ray absorptiometry, DXA (Lunar iDXA, GE Healthcare, IL, USA) for no-entry measurement to determine fat percentage
bone mineral density test | every 6 weeks
  Use dual-energy X-ray absorptiometry, DXA (Lunar iDXA, GE Healthcare, IL, USA) for no-entry measurement to determine bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chang Huang, Ph.D, Principal Investigator — PI
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Lee MC, Tu YT, Lee CC, Tsai SC, Hsu HY, Tsai TY, Liu TH, Young SL, Lin JS, Huang CC. Lactobacillus plantarum TWK10 Improves Muscle Mass and Functional Performance in Frail Older Adults: A Randomized, Double-Blind Clinical Trial. Microorganisms. 2021 Jul 8;9(7):1466. doi: 10.3390/microorganisms9071466. PMID 34361902